CLINICAL TRIAL: NCT05742451
Title: Investigation of the Effect of Yoga on Balance, Reaction Time and Agility in Children With Attention Deficit and Hyperactivity Disorder: A Randomized Controlled Trial
Brief Title: Investigation of the Effect of Yoga on Balance, Reaction Time and Agility in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Cemre Bafralı, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANKARAMEDİPOLUBAFRALİ001
Record Dates: First submitted 2022-12-30; First posted 2023-02-24 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Yoga; ADHD; Balance; Children, Only
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The kids yoga was applied to the intervention group for 8 weeks, once a week (8 sessions), 40 minutes per session, by a yoga instructor occupational therapist.
  Interventions: Other: kids yoga
- Control group (No Intervention): The control group was evaluated at 8-week intervals.

INTERVENTIONS:
Other: kids yoga — The kids yoga was applied to the intervention group for 8 weeks, once a week (8 sessions), 40 minutes per session, by a yoga instructor occupational therapist.
  Kids yoga training included: 5-minute warm-up consisting of jogging, jumping, stretching, relaxation exercises; 20 minutes of asanas (positions) consisting of standing, sitting, prone, supine postures and pranayamas (breathing exercises) consisting of vigorous inspiration and expiration, slow and rhythmic alternating nostril breathing; 10-minute yogic games about balance, reaction time and agility; meditation with focus for 5 minutes with resuscitation techniques.
  Arms: intervention group

SUMMARY:
Purpose: To determine the effect of 8-week kids yoga training on balance, reaction time and agility on children diagnosed with attention deficit hyperactivity disorder (ADHD).

Method: A randomized controlled trial. The intervention (kids yoga) was an 8-week program administered to children attending a special education center by a yoga instructor occupational therapist. Outcomes included Pediatric Balance Scale, Bruininks-Oseretsky Motor Proficiency Test-Short Form, and Microgate Witty SEM System assessed at baseline and at the end of 8th week.

DETAILED DESCRIPTION:
Introduction According to the fifth revision of the diagnostic and statistical manual of mental disorders (DSM-5), attention deficit and hyperactivity disorder (ADHD) is a heterogeneoud disorder that causes behavioral problems in at least two domains of life, lasting at least 6 months. Behavioral disorders usually manifest themselves in the school period and are characterized by hyper-motor skills, increased distractibility and attention disorders, impulsivity, and psychosocial adjustment disorders.

It is known that many children with ADHD have impairments in executive functions such as working memory, attention, emotion regulation, and inhibitory control. In addition to the cognitive function problems that are widely known and frequently emphasized in the literature, it is known that children with ADHD also have difficulties in activities that require motor coordination, such as handwriting. Several studies have found that children with ADHD perform poorly on motor skills tests assessing fine and gross motor areas.

Cho et al. (2014) stated that 30-70% of children with ADHD have motor control problems and these problems cause problems in their neurobehavioral development. School-age children with motor problems may face many problems such as the desire to avoid physical activity, obesity, lack of concentration, low self-esteem, school performance and inadequacy in social relations. Motor impairment, which causes problems with cycling, dressing, tying shoelaces and/or writing, may cause problems in children's social participation, peer relationships, and adaptation in daily life. Therefore, early detection and intervention of motor delay can reduce feelings of inadequacy, depression, frustration, and anxiety in children with ADHD and prevent long-term negative effects on social development and academic achievement.

The most commonly used treatment options for ADHD are pharmacological and psychosocial interventions. Parents may not prefer pharmacological methods because of their stimulating effect on the general health of their children. It is known that the effects of behavioral interventions cannot be generalized to non-target environments and behaviors. Considering these limitations, there is a trend towards different complementary methods for the treatment of ADHD. Among the complementary treatment options, there are methods such as meditation, yoga, massage, homeopathy, acupuncture, neurofeedback, nutritional supplements, and few foods diet.

In recent years, yoga programs for children have been widely used as a mind-body supplement and alternative medicine intervention to improve physical and mental health conditions, as the benefits of yoga practice in promoting general health are recognized. Yoga has many comprehensive types, and child yoga, one of them, is a fairly new type of yoga that can increase children's mental focus by providing mind, soul and body awareness, improve their enjoyment of life, social relationships, self-esteem and self-confidence levels. Kids yoga consists of compositions such as games, stories, postures, breathing exercises, imitations of living things in nature, memory games. While physical exercises (asanas) can increase the physical flexibility, coordination and strength, breathing practices and meditation are used to increase awareness and reduce anxiety and improve children's quality of life. Other beneficial effects include reduction of blood pressure, and improvements in endurance, mood, and metabolic regulation.

Yoga practiced in childhood mainly improves balance as well as proper postural alignment, musculoskeletal strength and endurance. In addition, the literature suggests that yoga training can improve motor planning, execution, reaction time, and agility. Studies conducted in many parts of the world have revealed the results on the effects of yoga in children, and various studies are carried out on the effect of yoga on short-term heart rate variability in children with autism, physical fitness in school-aged asthmatic children, psychomotor skills in mentally retarded children, and quality of life in children with hemophilia. In addition, there are studies on the effects of yoga on impulsivity, hyperactivity, attention and behaviors, executive functions and cognitive motor functions in children with ADHD. Yoga remains an investigational therapy, but more research is needed on its possible uses for this population. In this study, it was aimed to examine the effect of yoga on balance, reaction time and agility in children with ADHD.

Methods Study Design The present investigation is a cross-sectional study planned to examine the effect of yoga on balance, reaction time and agility in children with ADHD. An 8-week randomized controlled trial design following Consolidated Standards of Reporting Trials (CONSORT) recommendations was used in the study.

The study was carried out in accordance with the Declaration of Helsinki and was approved by the Ethics Committee of Non-Invasive Clinical Researches of Hacı Bektaş Veli University (No. 2100082713).

After the power analysis using G*Power version 3.1.9.4 software, it was calculated that 16 individuals with ADHD should be included in the study with a 5% type 1 error rate to reach 0.80 power. The minimum estimated sample was 15 participants, allowing for an estimated 15% dropout at follow-up.

Individuals were randomly divided into the intervention and control groups using computer-assisted online randomization application and simple randomization method in equal probability and in equal numbers, and kids yoga was applied to the intervention group. Participants were randomly numbered from 1 to 20, and the randomization of numbers under kids yoga (n=10) and control groups (n=10), without repeating the same number, using the online randomization application at https://www.randomizer.org/ appointed with. A total of 20 children were recruited and agreed to participate in the study. Because the individuals in the control group give education a rest, 3 participants left the study voluntarily.

The research team consisted of an occupational therapist who was blinded to the group distribution for assessments, an occupational therapist with a certificate of yoga training who conducted the yoga sessions, and physiotherapist and occupational therapist researchers who analyzed the evaluation results. The data were collected at 2 time points (baseline [April 2022] and post-test [June 2022]).

Participants The children who were diagnosed with ADHD by a child and adolescent psychiatrist according to DSM-V diagnostic criteria and were educated at Ankara Special Education Center were included in the study.

Inclusion criteria for the study were (1) the participants were between the ages of 6-10 and (2) received an occupational therapy treatment program. Exclusion criteria were (1) participants had a different diagnosis such as autism spectrum disorder, asperger's syndrome, pervasive developmental disorder, (2) had an additional psychiatric problem, (3) had a serious medical condition (for example, severe cerebral palsy) or intellectual disability (IQ < 70), (3) sought specialist help for sleep problems was determined as having a positive screening test for obstructive sleep apnea and (4) had excessive behavioral disorders incompatible with group participation.

Children who agreed to participate and met the inclusion criteria and their parents/guardians were informed about the aims of the study and their written informed consent was obtained.

Interventions The kids yoga was applied to the intervention group for 8 weeks, once a week (8 sessions), 40 minutes per session, by a yoga instructor occupational therapist.

Kids yoga training included: 5-minute warm-up consisting of jogging, jumping, stretching, relaxation exercises; 20 minutes of asanas (positions) consisting of standing, sitting, prone, supine postures and pranayamas (breathing exercises) consisting of vigorous inspiration and expiration, slow and rhythmic alternating nostril breathing; 10-minute yogic games about balance, reaction time and agility; meditation with focus for 5 minutes with resuscitation techniques.

Instruments Sociodemographic Information Form The sociodemographic information of the children was recorded in the information form. In the form, information such as date of birth, age, gender, school class, number of siblings, and parental marital status were obtained from the families of the children.

Pediatric Balance Scale (PBS) The Pediatric Balance Scale is an assessment that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points. The scale consists of sitting to standing, standing to sitting, transfers, standing unsupported, sitting unsupported, standing with eyes closed, standing with feet together, standing with one foot in front, standing on one foot, turning 360 degrees, turning to look behind, retrieving object from floor, placing alternate foot on stool, reaching forward with outstretched arm. In the study; ın the pedıatrıc balance scale standing with one foot in front, standing on one foot, turning 360 degrees, and placing alternate foot on stool sub-scales was applıed.

Bruininks-Oseretsky Test of Motor Proficiency-Short Form (BOT-SF) BOT-SF, which was developed to measure the motor functions of individuals between the ages of 4-21, is applied to the participants individually. The test materials, consisting of eight subtests and a total of 46 items, are a comprehensive motor proficiency indicator and measure both gross and fine motor skills.

BOT-SF materials are designed to attract children's attention, provide a uniform application opportunity, and facilitate application and evaluation. It consists of eight domains: running speed and agility, balance, bilateral coordination, endurance, arm-hand coordination, reaction speed, visual motor control, arm speed and manual dexterity. The highest score is 243 points. In our study, the response speed, running speed and agility sub-parameters of BOT-SF were used. In the BOT-SF running speed and agility sub-parameters, the score corresponding to the time in the distance run was recorded.

Microgate Witty SEM System The reaction time was recorded using the photocell system MICROGATE. The Witty SEM diagnostic system consists of eight photocells arranged in rows on a mat, 10 cm apart. Participants are asked to react as quickly as possible with their dominant hand to the green photocells that light up 20 times in sequence. In this test, visual stimuli are created immediately after each response. The best overall reaction time is recorded after two trials.

Statistical Analyses Statistical analyses were performed using SPSS software version 22. The variables were investigated using visual (histograms, probability plots) and analytical (Kolmogorov Simirnov/Shapiro Wilk test) methods to determine whether or not they are normally distributed. Descriptive analyses were presented using medians and interquartile ranges (IQR) for the non-normally distributed and ordinal variables. Since the data of children's age, balance scores, agility scores and reaction speed scores were not normally distributed, non-parametric tests were conducted to compare these parameters. The Mann-Whitney U test was used for pairwise comparisons for the intervention group and the control group. Wilcoxon Signed Rank Test was used to analyze pre- and post-measures for all variables. An overall 5% type-I error level was used to infer statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* The participants were between the ages of 6-10
* Received an occupational therapy treatment program

Exclusion Criteria:

* Participants had a different diagnosis such as autism spectrum disorder, asperger's syndrome, pervasive developmental disorder.
* Participants had an additional psychiatric problem
* Participants had a serious medical condition (for example, severe cerebral palsy) or intellectual disability (IQ < 70) sought specialist help for sleep problems was determined as having a positive screening test for obstructive sleep apnea.
* Participants had excessive behavioral disorders incompatible with group participation.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale (PBS) | 20 minutes
  The Pediatric Balance Scale is an assessment that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points. The scale consists of sitting to standing, standing to sitting, transfers, standing unsupported, sitting unsupported, standing with eyes closed, standing with feet together, standing with one foot in front, standing on one foot, turning 360 degrees, turning to look behind, retrieving object from floor, placing alternate foot on stool, reaching forward with outstretched arm. In the study; ın the pedıatrıc balance scale standing with one foot in front, standing on one foot, turning 360 degrees, and placing alternate foot on stool sub-scales was applıed.

SECONDARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency-Short Form (BOT-SF) | 20 minutes
  BOT-SF, which was developed to measure the motor functions of individuals between the ages of 4-21, is applied to the participants individually. The test materials, consisting of eight subtests and a total of 46 items, are a comprehensive motor proficiency indicator and measure both gross and fine motor skills.
  BOT-SF materials are designed to attract children's attention, provide a uniform application opportunity, and facilitate application and evaluation. It consists of eight domains: running speed and agility, balance, bilateral coordination, endurance, arm-hand coordination, reaction speed, visual motor control, arm speed and manual dexterity. The highest score is 243 points. In our study, the response speed, running speed and agility sub-parameters of BOT-SF were used. In the BOT-SF running speed and agility sub-parameters, the score corresponding to the time in the distance run was recorded

OTHER OUTCOMES:
Microgate Witty SEM System | 5 minutes
  The reaction time was recorded using the photocell system MICROGATE. The Witty SEM diagnostic system consists of eight photocells arranged in rows on a mat, 10 cm apart. Participants are asked to react as quickly as possible with their dominant hand to the green photocells that light up 20 times in sequence. In this test, visual stimuli are created immediately after each response. The best overall reaction time is recorded after two trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Cemre Bafralı, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No